CLINICAL TRIAL: NCT01123083
Title: Durable-Response Therapy Evaluation For Early- or New-Onset Type 1 Diabetes
Brief Title: Trial of Otelixizumab for Adolescents and Adults With Newly Diagnosed Type 1 Diabetes Mellitus (Autoimmune): DEFEND-2
Acronym: DEFEND-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115494; TRX4018 (Other: Tolerx)
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: new onset type 1 diabetes; juvenile diabetes; T1DM; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — otelixizumab; Antibodies, Monoclonal; Muromonab-CD3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- otelixizumab (Experimental): otelixizumab
  Interventions: Biological: Otelixizumab
- placebo (Placebo Comparator): placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Otelixizumab — infusion
  Other Names: ChAglyCD3; TRX4; monoclonal antibody; anti-CD3
  Arms: otelixizumab
Biological: Placebo — Infusion
  Arms: placebo

SUMMARY:
DEFEND-2 is a Phase 3 confirmatory study for the Phase 3 DEFEND-1 study. The study objective is to find out if an 8-day series of otelixizumab infusions leads to greater improvement in insulin secretion as compared with placebo. Insulin secretion will be assessed using mixed meal-stimulated C-peptide.

Subjects will be assigned to receive either otelixizumab or placebo at a ratio of 2:1 (2/3 otelixizumab, 1/3 placebo). These study agents will be administered as an addition to insulin, diet, and other standard of care treatments.

DETAILED DESCRIPTION:
The following visits are required:

* Screening Visits: 2 to 3 appointments will be conducted to determine eligibility. At 2 of these visits participants will drink a liquid meal and have blood tests done over the post-meal period. Participants will also be required to wear a continuous glucose monitor for a short period of time.
* Dosing Visits: 8 outpatient visits on consecutive days, each lasting about 2-4 hours.
* Follow-up Visits: weekly for the first month, then every 2 weeks for 3 months, followed by monthly visits through 1 year. There will be 3 visits in the second year.
* The total duration of the study is 2 years.
* Glucose test strips and glucose monitors will be provided to participants for the duration of the study. Frequent glycemic monitoring will occur through lab testing and blood glucose self-monitoring to help facilitate tight glycemic control in all subjects. Subjects will be asked to intermittently record their insulin doses using a telephone or web based system and continuous glucose monitoring will be performed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-17
* Diagnosis of diabetes mellitus, consistent with ADA criteria
* No more than 90 days between diagnosis and administration of study compounds
* Requires insulin for type 1 diabetes mellitus, or has required insulin at some time between diagnosis and administration of study compounds. In Canada, has to be using insulin at the time of dosing.
* Stimulated C-peptide level greater than 0.20 nmol/L and less than or equal to 3.50 nmol/L
* Positive for one or more of the autoantibodies typically associated with T1DM: antibody to glutamic acid decarboxylase (anti-GAD); antibody to protein tyrosine phosphatase-like protein (anti-IA-2); zinc transporter autoantibodies (ZNT8); insulin autoantibodies (IAA). A subject who is positive for insulin autoantibodies (IAA) and negative for the other autoantibodies will only be eligible if the subject has used insulin for less than 7 days total.

Exclusion Criteria:

•Other, significant medical conditions based on the study doctor's evaluation

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2012-03-09 (Actual); Study Completion 2012-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Keymeulen B, Vandemeulebroucke E, Ziegler AG, Mathieu C, Kaufman L, Hale G, Gorus F, Goldman M, Walter M, Candon S, Schandene L, Crenier L, De Block C, Seigneurin JM, De Pauw P, Pierard D, Weets I, Rebello P, Bird P, Berrie E, Frewin M, Waldmann H, Bach JF, Pipeleers D, Chatenoud L. Insulin needs after CD3-antibody therapy in new-onset type 1 diabetes. N Engl J Med. 2005 Jun 23;352(25):2598-608. doi: 10.1056/NEJMoa043980. PMID 15972866
- [Background] Keymeulen B, Walter M, Mathieu C, Kaufman L, Gorus F, Hilbrands R, Vandemeulebroucke E, Van de Velde U, Crenier L, De Block C, Candon S, Waldmann H, Ziegler AG, Chatenoud L, Pipeleers D. Four-year metabolic outcome of a randomised controlled CD3-antibody trial in recent-onset type 1 diabetic patients depends on their age and baseline residual beta cell mass. Diabetologia. 2010 Apr;53(4):614-23. doi: 10.1007/s00125-009-1644-9. Epub 2010 Jan 14. PMID 20225393
- [Background] You S, Candon S, Kuhn C, Bach JF, Chatenoud L. CD3 antibodies as unique tools to restore self-tolerance in established autoimmunity their mode of action and clinical application in type 1 diabetes. Adv Immunol. 2008;100:13-37. doi: 10.1016/S0065-2776(08)00802-X. No abstract available. PMID 19111162
- See also: Website containing information regarding the DEFEND-2 trial — http://www.defendagainstdiabetes.com
- Available data/document: Clinical Study Report: 115494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 73 centers in 10 countries (Belgium, Canada, Germany, Denmark, Spain, Finland, United Kingdom, Italy, Sweden, and United States of America) from 17 May 2010 to 09 March 2012.
Pre-assignment Details: A total of 179 participants (125 adults and 54 adolescents) were randomized in this study and included in safety and intent-to-treat (ITT) population.
Groups:
- Placebo: Eligible participants received Placebo matching otelixizumab 3.1 milligrams (mg) as intravenous (IV) infusion, with each infusion given over a 30-minute period. Participants received a series of 8 infusions, 1 infusion per day over 8 consecutive days.
- Otelixizumab: Eligible participants received otelixizumab 3.1 mg as IV infusion, with each infusion given over a 30-minute period. Participants received a series of 8 infusions, 1 infusion per day over 8 consecutive days.
Period: Overall Study
Arm/Group | Placebo | Otelixizumab
Started | 61 | 118
Completed | 50 | 103
Not Completed | 11 | 15
Not completed — Investigator recommendation | 1 | 1
Not completed — Administrative reasons | 0 | 4
Not completed — Lost to Follow-up | 2 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Withdrew for another reason not covered | 0 | 1
Not completed — Participant/legal representative request | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants received Placebo matching otelixizumab 3.1 mg as IV infusion, with each infusion given over a 30-minute period. Participants received a series of 8 infusions, 1 infusion per day over 8 consecutive days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Otelixizumab | Total
Number analyzed (Participants) | 61 | 118 | 179
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.5 (8.22) | 23.6 (8.34) | 23.2 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 50 | 74
  Male | 37 | 68 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 54 | 111 | 165
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 2 Hour Mixed Meal-stimulated C-peptide Area Under Curve (AUC) (Normalized for 120-minute Time Interval) at Month 12
Description: C-peptide is a protein that shows how much insulin the body is producing. For 3 days before the mixed meal tolerance test participants were asked to eat a balanced diet. The test was performed only when the finger-stick blood glucose level was above 70 mg per deciliter (mg/dL) and no higher than 200 mg/dL. Mixed meal-stimulated C-peptide AUC was the area under the C-peptide/time curve from time 0 to 120-minutes, calculated using the trapezoidal rule. This AUC was normalized for time interval by dividing it by 120-minutes (the number of minutes over which it was determined), and was adjusted by inclusion of Baseline C-peptide AUC as a covariate in the analysis. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the value at Month 12 from the Baseline value.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population consisted of all participants who were randomized and received any part of at least 1 infusion of study drug. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: nanomoles per liter
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 45 | 96
nanomoles per liter | -0.14 (0.036) | -0.23 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Test type: Superiority or Other; p = 0.051, Repeated Measures Mixed Effects Model; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.17 to 0.00] — Estimated treatment group difference, adjusted for age, region and Baseline C-peptide AUC. Confidence Interval, not adjusted for multiple comparisons

2. Secondary Outcome: Change From Baseline in 2 Hour Mixed Meal-stimulated C-peptide AUC (Normalized for 120-minute Time Interval) at Week 12 and 6 Months
Description: C-peptide is a protein that shows how much insulin the body is producing. For 3 days before the mixed meal tolerance test participants were asked to eat a balanced diet. The test was performed only when the finger-stick blood glucose level was above 70 mg/dL and no higher than 200 mg/dL. Mixed meal-stimulated C-peptide AUC was the area under the C-peptide/time curve from time 0 to 120-minutes, calculated using the trapezoidal rule. This AUC was normalized for time interval by dividing it by 120-minutes (the number of minutes over which it was determined), and was adjusted by inclusion of Baseline C-peptide AUC as a covariate in the analysis. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post Baseline value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 12, Month 6
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: nanomoles per liter
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
nanomoles per liter
  Week 12: number analyzed (Participants) | 55 | 105
  Week 12 | 0.05 (0.031) | -0.05 (0.023)
  Month 6: number analyzed (Participants) | 50 | 99
  Month 6 | -0.04 (0.037) | -0.10 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Week 12; Test type: Superiority or Other; p = 0.022, Repeated Measures Mixed Effects Model; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.18 to -0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Month 6; Test type: Superiority or Other; p = 0.191, Repeated Measures Mixed Effects Model; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.15 to 0.03] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Stimulated C-Peptide Mean AUC at Week 12, Month 6, 12 and 18
Description: as for outcome 2
Time Frame: Baseline (Day 1) and Week 12, Month 6, 12, 18
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
nanomoles per liter
  Week 12: number analyzed (Participants) | 55 | 105
  Week 12 | 0.0519 (0.24430) | -0.0472 (0.23394)
  Month 6: number analyzed (Participants) | 50 | 99
  Month 6 | -0.0455 (0.23802) | -0.0945 (0.29151)
  Month 12: number analyzed (Participants) | 45 | 96
  Month 12 | -0.1236 (0.24362) | -0.2331 (0.30537)
  Month 18: number analyzed (Participants) | 2 | 4
  Month 18 | -0.4125 (0.17059) | 0.0502 (0.25597)

4. Secondary Outcome: Number of Participants With Responder Status
Description: A participant was considered a responder when, at the given time point, the participant had: glycosylated hemoglobin (HbA1c) less than or equal to 6.5 percent and mean daily insulin use less than 0.5 international unit per kilogram per day (IU/kg/day) over 7 consecutive days during the 2 weeks preceding the visit.
Time Frame: Month 3, 6 and 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
Participants
  Week 12: number analyzed (Participants) | 41 | 68
  Week 12 | 19 | 42
  Month 6: number analyzed (Participants) | 35 | 61
  Month 6 | 11 | 26
  Month 12: number analyzed (Participants) | 27 | 54
  Month 12 | 10 | 23
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Week 12; Test type: Superiority or Other; p = 0.912, GEE Model; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.50 to 3.37] — Estimated treatment group difference, adjusted for age, region and Baseline HbA1c/Insulin Use Response. Confidence Interval, not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Month 6; Test type: Superiority or Other; p = 0.912, GEE Model; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.37 to 2.42] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Otelixizumab; Month 12; Test type: Superiority or Other; p = 0.412, GEE Model; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.54 to 4.52] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Mean Daily Insulin Use Over 7 Consecutive Days During the 2 Weeks Prior to the Assessment
Description: Mean daily insulin use over 7 consecutive days during the 2 weeks preceding each key visit was calculated as the mean of the values of amount of insulin used per day on each of the 7 consecutive days. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post Baseline value from the Baseline value.
Time Frame: Baseline (Day 1) and Month 3, 6, 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: International unit per kilogram (IU/kg)
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
International unit per kilogram (IU/kg)
  Week 12: number analyzed (Participants) | 35 | 55
  Week 12 | -0.04 (0.020) | -0.08 (0.016)
  Month 6: number analyzed (Participants) | 33 | 55
  Month 6 | 0.01 (0.027) | -0.04 (0.021)
  Month 12: number analyzed (Participants) | 26 | 45
  Month 12 | 0.01 (0.036) | 0.05 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Week 12; Test type: Superiority or Other; p = 0.210, Repeated Measures Mixed Effects Model; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.08 to 0.02] — Estimated treatment group difference, adjusted for age, region and Baseline Mean Daily Insulin Use. Confidence Interval, not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Month 6; Test type: Superiority or Other; p = 0.210, Repeated Measures Mixed Effects Model; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.11 to 0.02] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Otelixizumab; Month 12; Test type: Superiority or Other; p = 0.402, Repeated Measures Mixed Effects Model; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.05 to 0.13] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in HbA1c Levels Over 7 Consecutive Days During the 2 Weeks Prior to the Assessment
Description: HbA1c level was recorded at Baseline, Month 3, 6 and 12. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post Baseline value from the Baseline value.
Time Frame: Baseline (Day 1) and Month 3, 6, 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
Percentage of HbA1c
  Week 12: number analyzed (Participants) | 58 | 109
  Week 12 | -0.82 (0.140) | -1.01 (0.101)
  Month 6: number analyzed (Participants) | 54 | 94
  Month 6 | -0.65 (0.185) | -0.65 (0.134)
  Month 12: number analyzed (Participants) | 48 | 99
  Month 12 | -0.61 (0.188) | -0.47 (0.133)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Week 12; Test type: Superiority or Other; p = 0.582, Repeated Measures Mixed Effects Model; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.52 to 0.16] — Estimated treatment group difference, adjusted for age, region and baseline HbA1c. Confidence Interval, not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Month 6; Test type: Superiority or Other; p = 0.987, Repeated Measures Mixed Effects Model; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.46 to 0.45] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Otelixizumab; Month 12; Test type: Superiority or Other; p = 0.572, Repeated Measures Mixed Effects Model; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.33 to 0.59] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Average Number of Severe Hypoglycemic Events and Documented Symptomatic Hypoglycemic Events From Baseline to Month 12
Description: Severe hypoglycemia was considered as an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. Plasma glucose measurements may not be available during such an event, but neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. Documented symptomatic hypoglycemia was considered as an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration less than or equal to 70 mg/dL and it was collected in (1) eCRF using two forms - for single event and for mutiple events, and (2) the IVRS system. The numbers of participant-reported hypoglycemic events per participant of severe hypoglycemia and documented symptomatic hypoglycemia have been reported.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population.
Measure: Number; unit: Events
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
Events
  Severe hypoglycemia | 33 | 11
  Documented symptomatic hypoglycemia from IVRS | 429 | 690
  Documented symptomatic hypoglycemia from eCRF | 822 | 1300

8. Secondary Outcome: Percentage of Participants With Change From Baseline in Severe Hypoglycemic Events and Documented Symptomatic Hypoglycemic Events at Month 12
Description: Severe hypoglycemia was considered as an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. Plasma glucose measurements may not be available during such an event, but neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. Documented symptomatic hypoglycemia was considered as an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration less than or equal to 70 mg/dL and it was collected in (1) eCRF using two forms - for single event and for mutiple events, and (2) the IVRS system. The percentage of participant with incidence of severe hypoglycemia and documented symptomatic hypoglycemia have been reported.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
Percentage of participants
  Severe hypoglycemia | 11.5 | 5.9
  Documented symptomatic hypoglycemia from IVRS | 36.1 | 28.8
  Documented symptomatic hypoglycemia from eCRF | 45.9 | 43.2

9. Secondary Outcome: Composite Rank Sum: HbA1c and Exogenous Insulin Use at 6 and 12 Months
Description: O'Brien mean rank analyses was performed on a two-part composite of the Baseline-adjusted HbA1c level and the Baseline-adjusted mean total daily insulin use per kg body weight in the otelixizumab group compared with the placebo group at Months 6 and 12. Baseline adjustment was used to reduce the potential impact of imbalances in Baseline levels between treatment groups on the treatment comparisons at later time points. For the O'Brien mean rank analysis at a particular time point, adjusted HbA1c values (for both treatment groups together) and adjusted mean daily insulin use values was ranked from smallest to largest. For each participant, the HbA1c and insulin use ranks were added together, producing a composite rank. A treatment comparison test was then performed on the composite ranks. If otelixizumab treatment was effective on this composite endpoint, then the mean of the ranks sum in the otelixizumab group was smaller than the mean of the ranks sum in the placebo group.
Time Frame: Month 6 and 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Rank
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
Rank
  Month 6: number analyzed (Participants) | 28 | 48
  Month 6 | 119 (48.4) | 110 (49.8)
  Month 12: number analyzed (Participants) | 23 | 45
  Month 12 | 96 (51.2) | 110 (55.3)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Month 6; Test type: Superiority or Other; p = 0.452, Hochberg-adjusted p-value
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Month 12; Test type: Superiority or Other; p = 0.452, Hochberg-adjusted p-value

10. Secondary Outcome: Composite Rank Sum: C-Peptide AUC, HbA1c and Exogenous Insulin Use at 6 and 12 Months
Description: O'Brien analyses was performed on a three-part composite of HbA1c level, C-peptide AUC, and mean daily insulin use in the otelixizumab group compared with the placebo group at Months 6 and 12. The three variables was adjusted for Baseline values. Baseline adjustment was used to reduce the potential impact of imbalances in Baseline levels between treatment groups on the treatment comparisons at later time points. HbA1c and insulin use was ranked from smallest to largest, and C-peptide AUC was ranked from largest to smallest. If otelixizumab treatment was effective on the composite endpoint, then the mean of the ranks sum in the otelixizumab group was smaller than the mean of the ranks sum in the placebo group.
Time Frame: Month 6 and 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Rank
Arm/Group | Placebo | Otelixizumab
Number analyzed (Participants) | 61 | 118
Rank
  Month 6: number analyzed (Participants) | 26 | 48
  Month 6 | 206 (48.6) | 186 (41.6)
  Month 12: number analyzed (Participants) | 23 | 42
  Month 12 | 180 (42.5) | 170 (46.0)
Statistical Analysis 1: Comparison: Placebo vs Otelixizumab; Month 6; Test type: Superiority or Other; p = 0.123, Hochberg-adjusted p-value
Statistical Analysis 2: Comparison: Placebo vs Otelixizumab; Month 12; Test type: Superiority or Other; p = 0.373, Hochberg-adjusted p-value

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from dosing Days 1 to 8 and until study withdrawal.
Description: Safety population consisted of all participants for whom there was evidence that they received any part of at least 1 infusion of study drug.
Arm/Group | Placebo | Otelixizumab
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/118
Serious Adverse Events (participants affected / at risk) | 4/61 | 11/118
Other Adverse Events (participants affected / at risk) | 50/61 | 108/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | Otelixizumab (N=118)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | Otelixizumab (N=118)
Headache (Nervous system disorders) | 34 | 92
Dizziness (Nervous system disorders) | 4 | 12
Nasopharyngitis (Infections and infestations) | 15 | 37
Upper respiratory tract infection (Infections and infestations) | 16 | 9
Sinusitis (Infections and infestations) | 7 | 3
Influenza (Infections and infestations) | 0 | 9
Pharyngitis streptococcal (Infections and infestations) | 0 | 6
Urinary tract infection (Infections and infestations) | 0 | 6
Nausea (Gastrointestinal disorders) | 16 | 38
Vomiting (Gastrointestinal disorders) | 2 | 19
Abdominal pain (Gastrointestinal disorders) | 5 | 11
Diarrhoea (Gastrointestinal disorders) | 1 | 11
Abdominal pain upper (Gastrointestinal disorders) | 1 | 6
Fatigue (General disorders) | 11 | 28
Pyrexia (General disorders) | 2 | 21
Chills (General disorders) | 3 | 16
Malaise (General disorders) | 4 | 4
Infusion site erythema (General disorders) | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.